CLINICAL TRIAL: NCT06749860
Title: Disitamab Vedotin in Combination with Tislelizumab and Bevacizumab in a Phase II Clinical Study of Locally Advanced or Metastatic Non-small Cell Lung Cancer with HER2 Mutation/amplification/expression
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Chunxia Su, Director of the Clinical Research Center, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023LY0833
Record Dates: First submitted 2024-12-12; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — disitamab vedotin; tislelizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- treated (Experimental): Patients with locally advanced or metastatic NSCLC who have received prior ≥1-line systemic therapy
  Interventions: Drug: Disitamab Vedotin + tislelizumab + bevacizumab
- treatment-navie (Experimental): Patients with locally advanced or metastatic NSCLC who have not received prior systemic therapy
  Interventions: Drug: Disitamab Vedotin + tislelizumab + bevacizumab

INTERVENTIONS:
Drug: Disitamab Vedotin + tislelizumab + bevacizumab — Disitamab Vedotin, dosing regimen: 2.0 mg/kg, intravenous infusion, infusion should be about 30-90 minutes (usually about 60 minutes), every 21 days a cycle, the first day of administration, continuous use.
  Tislelizumab, dosing regimen: 200 mg administered by intravenous infusion every 21 days in a cycle on the first day, continuous.
  Bevacizumab, dosing regimen; 7.5 mg/kg administered by intravenous infusion every 21 days in a cycle on the first day of continuous use.

SUMMARY:
The goal of this clinical trial is to learn ifDisitamab Vedotin in combination with tislelizumab and bevacizumab can treat in locally advanced or metastatic non-small cell lung cancer patients with HER2 mutation/amplification/expression. The main questions it aims to answer are:

1. objective response rate;
2. Progression-Free Survival;
3. Overall Survival;
4. Disease Control Rate;
5. Duration of Response.

ELIGIBILITY:
Inclusion Criteria:

1. Prior to the implementation of any trial-related procedures, written informed consent must be obtained;
2. Aged >= 18 years;
3. Patients with locally advanced (Stage III B/III C), metastatic, or recurrent (Stage IV) non-small cell lung cancer (NSCLC) confirmed histologically or cytologically, who are ineligible for surgical intervention and cannot undergo curative radiochemotherapy, as per the 8th edition TNM staging classification of the International Association for the Study of Lung Cancer and the American Joint Committee on Cancer;
4. Provision of archived tumor tissue or tissue obtained during screening biopsy for biomarker testing, including PD-L1 expression, HER2 mutation status, etc.;
5. HER2 mutation, amplification, or HER2 expression (IHC 1+, 2+, or 3+);
6. Investigator confirmation of at least one measurable lesion according to RECIST 1.1 criteria;
7. Cohort I: Patients who have received prior ≥1 line of systemic therapy or HER2 tyrosine kinase inhibitors such as afatinib, pyrotinib, or pozitinib. Cohort II: No prior receipt of any systemic anti-tumor therapy for advanced/metastatic disease; For patients who have previously received platinum-containing adjuvant/radiotherapy, neoadjuvant/radiotherapy, or radical chemoradiotherapy for advanced disease, disease progression occurs >6 months after the end of the last treatment, may participate in this study;
8. Expected life expectancy >= 3 months;
9. ECOG PS 0-1;
10. Adequate hematologic function, defined as an absolute neutrophil count >= 1.5×10^9/L, platelet count >= 100×10^9/L, hemoglobin >= 90g/L (without a history of blood transfusion in the past 7 days);
11. Adequate liver function, defined as total bilirubin level <= 1.5 times the upper limit of normal (ULN) and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels <= 2.5 times ULN for all patients, or for patients with liver metastasis, AST and ALT levels <= 5 times ULN;
12. Adequate renal function, defined as serum creatinine <= 1.5 times ULN;
13. Adequate coagulation function, defined as international normalized ratio (INR) or prothrombin time (PT) <= 1.5 times ULN; if a subject is on anticoagulant therapy, INR/PT should be within the therapeutic range set by the anticoagulant;
14. Women of childbearing potential must undergo a pregnancy test within 7 days prior to the start of treatment, with negative results; and reliable contraception methods (such as intrauterine devices, oral contraceptives, and condoms) should be used during the trial and for 30 days after the end of the trial. Men of childbearing potential should use condoms for contraception during the trial and for 30 days after the end of the trial;
15. Willingness to comply with regular follow-up visits and adhere to trial requirements.

Exclusion Criteria:

1. Currently participating in interventional clinical research treatment;
2. Prior treatment with HER2 antibodies or antibody-drug conjugates;
3. Received traditional Chinese medicine or immunomodulatory drugs (such as thymopeptides, interferons, interleukins, etc.) with anti-tumor indications within the 2 weeks preceding the first dose;
4. Patients undergoing EGFR-TKI treatment require a 2-week washout period;
5. History of allergic reactions to any components of the investigational drug;
6. Presence of clinically significant active hemoptysis, active diverticulitis, intra-abdominal abscess, gastrointestinal obstruction, or peritoneal metastasis requiring clinical intervention;
7. Presence of clinically uncontrollable pleural effusion/ascites (patients not requiring drainage or with no significant increase in effusion for 3 days may be eligible);
8. Tumor compression of vital surrounding organs (such as the esophagus) accompanied by relevant symptoms, compression of the superior vena cava, or invasion of major mediastinal vessels, heart, etc.;
9. Severe complications such as a history of severe pulmonary or cardiac diseases; occurrence of any arterial thrombosis, embolism, or ischemia within 6 months prior to enrollment, including myocardial infarction, unstable angina, cerebrovascular accident, or transient ischemic attack. A history of deep vein thrombosis, pulmonary embolism, or any other serious thromboembolic event within the past 3 months before enrollment;
10. Known presence of brain metastases. Asymptomatic or stable patients with brain metastases, as judged by the investigator, may be eligible;
11. Received systemic corticosteroids (>10 mg/day prednisone or equivalent) or other systemic immunosuppressive agents (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, mercaptopurine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within the 2 weeks prior to enrollment. Local, ocular, intra-articular, intranasal, and inhaled corticosteroids are allowed;
12. History of autoimmune diseases, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vasculitis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis. Patients with autoimmune-related hypothyroidism receiving stable doses of thyroid hormone replacement therapy are eligible. Patients with controlled type 1 diabetes on stable insulin regimens are eligible;
13. Active systemic infections, including tuberculosis (clinically diagnosed based on medical history, physical examination, imaging findings, and routine TB examinations), hepatitis B (known positive for hepatitis B surface antigen [HBsAg] with HBV DNA >= 1000 cps/ml or its reference lower limit), hepatitis C, or human immunodeficiency virus (HIV antibody positive);
14. Known psychiatric disorders or substance abuse that may affect compliance with trial requirements;
15. Recent use of a sufficient dose of oral or non-oral anticoagulants or thrombolytic agents. Prophylactic use of anticoagulants is allowed;
16. History, diseases, treatments, or laboratory abnormalities that may interfere with trial results, hinder the subject's full participation in the study, or are deemed by the investigator to be against the subject's best interests in participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2024-02-02 (Actual); Primary Completion 2026-06-06 (Estimated); Study Completion 2027-06-06 (Estimated)

PRIMARY OUTCOMES:
objective response rate | up to 1 year
  It refers to the proportion of patients whose tumors shrink to a certain amount and remain for a certain period of time, including cases of complete response (CR) and partial response (PR).

SECONDARY OUTCOMES:
Progression-Free Survival | up to 1 year
  Refers to the time from the date of initiation of combination therapy to any objectively documented tumor progression or patient death (the last follow-up time for patients lost to follow-up; Patients who are still alive at the end of the study will be the end of follow-up at the end of the study).
Overall Survival | up to 1 year
  refers to the time from the start of combination therapy to the patient's death (the last follow-up time for patients who are lost to follow-up; Patients who are still alive at the end of the study will be the end of follow-up at the end of the study).
Disease Control Rate | 1 year
  Refers to the proportion of patients whose tumors shrink to a certain amount and remain for a certain period of time, including cases of complete response (CR), partial response (PR) and stable (SD).
Duration of Response | 1 year
  The duration of a patient's life from the first documented confirmed response (CR or PR) to the first documented disease progression (PD) or death due to any cause (whichever occurs first)

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No